CLINICAL TRIAL: NCT06781788
Title: I Want to Talk About Climate Change, But I Wish I Didn't Have to… A Descriptive Qualitative Study of an Intervention Combining Creative Arts and Philosophical Inquiry to Help Elementary School Students Cope With Climate Change Emotions
Brief Title: School-based Intervention to Address Climate Change Emotions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec a Montréal (Other)
Collaborators: Bishop's University (Other)
Responsible Party: Principal Investigator, Terra Léger-Goodes, Principal investigator, Université du Québec a Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 767-2023-1376-1
Record Dates: First submitted 2025-01-07; First posted 2025-01-17 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-01

CONDITIONS: Eco-anxiety
Keywords: Eco-anxiety in children; Creative arts intervention; Philosophical inquiry intervention; School-based intervention

STUDY DESIGN:
Intervention Model Description: The ORBIT model for intervention development is a framework developed by Czajkowski and colleagues (2015) in collaboration with the National Institute for Health. The model is a systematic approach that helps guide researchers through the various stages of intervention development, evaluation and implementation. The model emphasizes the iterative and dynamic nature of intervention development and evaluation. Phase 1b aims to refine the intervention to optimize it while retaining the components essential to its power to change, which corresponds to the first part of this framework. The data obtained in the previous phase are therefore taken into account to maximize the intervention's effectiveness. Among other things, qualitative methods to assess the acceptability of the intervention in the target population can be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Creative arts an philosophy inquiry intervention (Other): Participation in a seven-week school-based creative arts and philosophy inquiry intervention to talk about climate change emotions
  Interventions: Other: Making room for climate emotions in the classroom

INTERVENTIONS:
Other: Making room for climate emotions in the classroom — The "Making room for climate emotions in the classroom" program is designed to address emotions as students learn (formally or informally) about climate change. Each session features a drawing, photography, Lego sculpture, rock painting or collage/drawing workshop to address themes, explore emotions/feelings/experiences and initiate discussions on topics related to climate change.

SUMMARY:
The goal of this study was to qualitatively document the social validity of an intervention combining creative arts and philosophy inquiry and to examine its acceptability, the perceived goals, and perceived benefits for children's mental health and ability to cope with climate change from the perspective of one elemetary-school class students and their teacher.

The guiding research question was: How do children and their teacher perceive the acceptability, the goals and the benefits of the intervention? The participants were asked to participate in a seven-week creative arts and philosophical inquiry intervention. Once a week, a research assistant led a workshop using creative arts and group philosophical inquiry to discuss the topic of climate change and the emotions that can arise. Students participated in a brief individual interview after the intervention. The teacher also participated in an individual online interview.

ELIGIBILITY:
Inclusion Criteria:

* Elementary school students between the ages of 8 and 12 years old who's teacher accepted to participate in the study
* Elementary school teacher

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Social validity of the intervention | Immediately after the end of the intervention (at week 7)
  The social validity comprises of the perceived acceptability, goals and benefits of the intervention from participants' perspectives. It was measured using semi-structured interviews with open-ended questions to allow children and teachers to freely describe in detail their experience of the intervention. The interview guide was developed by the research team and piloted in previous research project to ensure that children understood the questions and that it allowed both positive and negative elements related to the intervention to emerge.

CONTACTS AND LOCATIONS:
Locations (1):
- Bishop's University, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analyzed during the current study are not publicly available due to the nature of qualitative data that might contain identifying information through the interview (e.g., speech slurs) but are available from the corresponding author upon reasonable request. The manuscript contains excerpts of the verbatim content that support each of the themes presented. Full data are not made available to ensure the confidentiality of the participants.

REFERENCES:
- [Derived] Leger-Goodes T, Herba CM, Piche J, Smith J, Ethier MA, Lefrancois D, Malboeuf-Hurtubise C. I want to talk about climate change, but I wish I didn't have to: A descriptive qualitative study of an intervention combining creative arts and philosophical inquiry to help elementary school students cope with climate change emotions. BMC Psychol. 2025 Dec 8;13(1):1339. doi: 10.1186/s40359-025-03589-w. PMID 41361496